CLINICAL TRIAL: NCT04229251
Title: Efficacy of Online Mindfulness-Based Intervention on Emerging Malaysian Chinese Adults With Attention Deficit/Hyperactivity Disorder: A Randomized Controlled Trial
Brief Title: Online Mindfulness-Based Intervention for ADHD
Acronym: iMBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universiti Tunku Abdul Rahman (Other)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Pheh Kai Shuen, Lecturer, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U/SERC/93/2019
Record Dates: First submitted 2019-12-29; First posted 2020-01-18 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-01

CONDITIONS: Attention-deficit Hyperactivity Disorder
Keywords: Mindfulness; Online intervention; Malaysia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Mindfulness-based Intervention (Experimental): iMBI will be delivered to participants in 8 online sessions, approximately 2 hours per session.
  Interventions: Behavioral: Online Mindfulness-based Intervention
- Online Introductory Psychology Program (Sham Comparator): An online introductory psychology courses will be delivered to participants in 8 online sessions, approximately 2 hours per session.
  Interventions: Behavioral: Online Introductory Psychology Program

INTERVENTIONS:
Behavioral: Online Mindfulness-based Intervention — The iMBI starts with psychoeducation about ADHD and defining mindfulness. Participants were then encouraged to discuss their experience of living with ADHD via a series of guided questions. Upon orientated to the program, the participants will be introduced to various topics of mindfulness and ADHD, as well as a wide range of in-session online mindfulness exercises. Offline assignments that correspond to each week's theme will be assigned to participants at the end of each session. Downloadable audio tracks for offline practices will be provided to the participants. Participants are expected to spend around 15 to 30 minutes each day to complete the weekly iMBI assignment.
  Other Names: iMBI
  Arms: Online Mindfulness-based Intervention
Behavioral: Online Introductory Psychology Program — The online introductory psychology program is a mass online open course program, providing comprehensive overview about psychology as an academic discipline. Each week, participants will be presented with approximately 2-hours pre-recorded lecture. Offline assignments that correspond to each week's theme will be assigned to participants at the end of each session.Downloadable handouts for revision will be provided to the participants. Participants are encouraged to spend around 15 to 30 minutes each day to complete the weekly assignment.
  Arms: Online Introductory Psychology Program

SUMMARY:
This study aims to evaluate the efficacies of an online mindfulness-based intervention for emerging adults with ADHD in Malaysia. The investigators hypothesized that online mindfulness-based intervention may improve ADHD symptoms and executive functions of emerging adults with ADHD.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a common neurodevelopmental disorder that often persist to adulthood. In Malaysia, the Chinese ethnic is having the highest prevalence rate of hyperactivity symptoms. Nevertheless, there are only limited evidence-based treatment options targeting the core symptoms of ADHD, as well as executive functions in adulthood. In addition, conventional psychotherapeutic approaches for adults with ADHD have found to be highly labor-intensive. Emerging adulthood is a distinct developmental stage of 18 - 29 years old, with unique challenges that rarely addressed in mental health system. Recently, mindfulness-based intervention appears to be a promising treatment for adults living with ADHD but it has not been evaluated among Malaysian emerging adults with ADHD. The investigators proposed a two-arm randomized controlled trial, comparing an eight-week online mindfulness-based intervention program with an online introductory psychology program. The outcomes include changes of inattention symptom, changes of hyperactivity-impulsivity symptom, and changes of executive functions from pretest to posttest, 1-month follow-up and 3-month follow-up. To investigators' best knowledge, this randomized controlled trial will be the first to test the efficacious of online mindfulness-based intervention for ADHD among emerging adults. It will provide evidence on the efficacious of online treatment for this often-overlooked population in the mental healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 29 years old.
* Diagnosis of ADHD.
* Completed at least six years of Chinese education.
* Participants taking psychotropic prescriptions will be allowed to participate, if they prescriptions were stable for at least 6 weeks prior to their participation in this study.

Exclusion Criteria:

* History or current presence of substance dependence, psychotic illness, bipolar disorder, personality disorders, conduct disorder, chronic suicidal, or self-injurious behaviour as reported in the Diagnostic Interview For Anxiety, Mood, Obsessive-Compulsive and Related Neuropsychiatric Disorders (DIAMOND).
* Non-verbal intellectual ability of percentile ranks 25 or below.
* Received cognitive-behavioural therapy (CBT) for ADHD or any form of mindfulness-based intervention in the past 2 years.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from pretest Inattention scores at posttest. | 8 weeks
  The ADHD Self-Report Scale (Inattention Subscale) is used in monitoring treatment response of Adult ADHD. The Inattention subscale scores range from 0 to 36, where higher scores indicate more severe levels of inattention.
Change from pretest Inattention scores at 1-month follow-up. | 12 weeks
  The ADHD Self-Report Scale (Inattention Subscale) is used in monitoring treatment response of Adult ADHD. The Inattention subscale scores range from 0 to 36, where higher scores indicate more severe levels of inattention.
Change from baseline Inattention scores at 3-month follow-up | 20 weeks
  The ADHD Self-Report Scale (Inattention Subscale) is used in monitoring treatment response of Adult ADHD. The Inattention subscale scores range from 0 to 36, where higher scores indicate more severe levels of inattention.
Change from pretest Hyperactivity-Impulsivity scores at posttest. | 8 weeks
  The ADHD Self-Report Scale (Hyperactivity-Impulsivity Subscale) is used in monitoring treatment response of Adult ADHD. The Hyperactivity-Impulsivity subscale scores range from 0 to 36, where higher scores indicate more severe levels of hyperactivity-impulsivity.
Change from pretest Hyperactivity-Impulsivity scores at 1-month follow-up. | 12 weeks
  The ADHD Self-Report Scale (Hyperactivity-Impulsivity Subscale) is used in monitoring treatment response of Adult ADHD. The Hyperactivity-Impulsivity subscale scores range from 0 to 36, where higher scores indicate more severe levels of hyperactivity-impulsivity.
Change from pretest Hyperactivity-Impulsivity scores at 3-month follow-up. | 20 weeks
  The ADHD Self-Report Scale (Hyperactivity-Impulsivity Subscale) is used in monitoring treatment response of Adult ADHD. The Hyperactivity-Impulsivity subscale scores range from 0 to 36, where higher scores indicate more severe levels of hyperactivity-impulsivity.
Change from pretest Executive Function Deficits scores at posttest. | 8 weeks
  The Adult Executive Functioning Inventory (ADEXI) is used in monitoring treatment response of Adult ADHD. The Executive Function Deficits subscale scores range from 14 to 70, where higher scores indicate more severe levels of executive function deficits.
Change from pretest Executive Function Deficits scores at 1-month follow-up. | 12 weeks
  The Adult Executive Functioning Inventory (ADEXI) is used in monitoring treatment response of Adult ADHD. The Executive Function Deficits subscale scores range from 14 to 70, where higher scores indicate more severe levels of executive function deficits.
Change from pretest Executive Function Deficits scores at 3-month follow-up. | 20 weeks
  The Adult Executive Functioning Inventory (ADEXI) is used in monitoring treatment response of Adult ADHD. The Executive Function Deficits subscale scores range from 14 to 70, where higher scores indicate more severe levels of executive function deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Shuen Pheh, MClinPsych, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Universiti Tunku Abdul Rahman, Kampar, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
All outcome measures data may be shared OSF Platform after the publications.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after December 2022.
Access Criteria: Data collected from this study, including de-identified individual participant data, will be made available upon publication to members of the scientific and medical community for non-commercial use only, upon email request to the corresponding author. The study protocol, statistical analysis plan, and informed consent forms are available on ClinicalTrials.gov.

REFERENCES:
- [Derived] Pheh KS, Tan KA, Ibrahim N, Sidik SM. Effectiveness of Online Mindfulness-Based Intervention (iMBI) on Inattention, Hyperactivity-Impulsivity, and Executive Functioning in College Emerging Adults with Attention-Deficit/Hyperactivity Disorder: A Study Protocol. Int J Environ Res Public Health. 2021 Jan 30;18(3):1257. doi: 10.3390/ijerph18031257. PMID 33573341